CLINICAL TRIAL: NCT06162689
Title: Do Risk Factors for Postpartum Psychosis Alter Offspring Outcomes in Middle Childhood
Brief Title: Psychiatry Research and Motherhood at 6 to 8 (PRAM-P@6to8)
Acronym: PRAM-P@6to8
Status: Enrolling by invitation | Type: Observational
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24.03.23 v1.0
Record Dates: First submitted 2023-03-27; First posted 2023-12-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Perinatal Psychiatry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples from adult participants and their children to assess salivary cortisol. Blood serum is collected from participants for the assessment of inflammatory markers and transcriptomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed Group: Women at risk of postpartum psychosis during pregnancy
- Unexposed Group: Women with no current or past history of psychiatric disorders during pregnancy

SUMMARY:
The goal of this observational study is to examine the relationship between severe perinatal maternal mental illness and stress reactivity and general development of children aged 6 to 8 years. Mothers were previously recruited and assessed during pregnancy and their babies were assessed at 6 days, 8 weeks and 12 months post delivery. This follow-up will assess the occurrence of any psychiatric episodes (e.g., depression, mania, psychosis) in the intervening period. Assessments of the children will include evaluation of their response to a mildly stressful procedure, as well as their physical, cognitive and social-emotional development, and their mental health. Possible factors that may moderate the relationship between the mother's perinatal mental health and the child's stress reactivity and development, including the home environment, adversity, parent-child interaction and maternal and paternal (or co-parent) mental health will also be assessed.

DETAILED DESCRIPTION:
The principle research question is "does maternal stress system in pregnant women at risk of postpartum psychosis modify stress reactivity in children aged 6 to 8"?.

The "stress system" the investigators are studying is the endocrine system known as the hypothalamic-pituitary-adrenal (HPA) axis. The investigators measured levels of hormones from this system in blood and saliva in a sample of women at risk and not at risk of postpartum psychosis during pregnancy and measured cortisol in the saliva of their babies, before and after a stressful experience at 6 days, 8 weeks and 12 months of age.

The investigators found that infants born to women at risk of postpartum psychosis (PP) who relapsed in the first 4 weeks post-delivery had altered HPA axis activity at 6 days post-birth, compared with infants born to women at risk who remained well in the postpartum period.

The investigators now plan to examine whether levels of mothers' stress hormones associated with risk of postpartum psychosis during pregnancy are also associated with longer-lasting children's cortisol stress reactivity and diurnal rhythm of cortisol during middle childhood (ages 6 to 8).

Genetic material will be extracted from the child's specimens to look at genes, epigenetics (DNA methylation) and changes in gene expression, specifically, changes in genes which might be relevant to the development of stress. Assessments of maternal endocrine and maternal and paternal / co-parent mood measures will be undertaken. Children's cortisol response to stress and cortisol diurnal rhythm will be carried out at ages 6 to 8 years, together with assessments of their growth, cognitive development, social-emotional functioning and mental health. The father or co-parent mental health, their relationship with the mother and their interaction/relationship with the child will also be measured to investigate whether these moderate any effects of maternal perinatal mental health on child development.

Prospective participants (n=72) were recruited in pregnancy, to take part in a study entitled "Risk factors of perinatal mental disorders: stress, electrophysiological and neuroimaging markers", also known as the Psychiatry Research and Motherhood - Psychosis (PRAM-P) study. Clinical assessments were undertaken in pregnancy and, following delivery, assessments of the infant and mother were undertaken at 6 days, 8 weeks and 12 months post delivery. At the final visit, 67 participants gave their written consent to be contacted at some time in the future to discuss the possibility of participating in a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the previous study (Risk factors of perinatal mental disorders: Stress, electrophysiological, and neuroimaging markers), who gave consent to be contacted again, together with their offspring, and the child's father/co-parent.

Exclusion Criteria:

* Women who participated in the previous study who refused consent to be contacted again.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study comprised 2 groups: women at risk of postpartum psychosis during pregnancy (exposed group) and women with no current or past history of psychiatric disorders (unexposed group).
  Cases were women at risk of postpartum psychosis because of a DSM-IV diagnosis of bipolar disorder, schizoaffective disorder or previous postpartum psychosis and controls were women who did not have a current or past history of psychiatric disorders. Clinical assessments were undertaken in the second and third trimesters of pregnancy and, following delivery, assessments of mother and infant were undertaken at 6 days, 8 weeks and 12 months post-delivery (n=72). At this stage, participants were asked to provide written consent to be contacted in the future about the possibility of taking part in a follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Child Salivary Cortisol | 6-8 years
  Child stress response - salivary cortisol: saliva samples will be collected before and after a mild stressor test: Cold Pressor Test (CPT) to assess stress reactivity.
Child Salivary Cortisol | 6-8 years
  Child stress response - salivary cortisol: saliva samples will be collected before and after a mild stress test: MacArthur Story Stem battery (MSSB) to asses stress reactivity

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children (4th Edition) (WISC-IV) | 6-8 years
  Child Cognitive Development
Wechsler Individual Achievement Test Second UK Edition (WIAT-II UK) | 6-8 years
  Child Cognitive Development
Dimensional Change Card Sort Test (DCCS) | 6-8 years
  Child Cognitive Development
Depression Self-Rating Scale (DSRS) | 6-8 years
  Child Mental Health
State-Trait Anxiety Inventory for Children (STAIC) | 6-8 years
  Child Mental Health
Strengths and Difficulties Questionnaire (SDQ) | 6-8 years
  Child emotional/behavioural symptoms and mental health, parent-report.
Development and Well-Being Assessment (DAWBA). | 6-8 years
  Child emotional/behavioural symptoms and mental health, parent-report.
Juvenile Victimization Questionnaire (JVQ) | 6-8 years
  Child social-relational risk factors, parent-report.
Traumatic Events Screening Inventory (TESI) | 6-8 years
  Child social-relational risk factors, parent-report.
Child Rearing Practices Report (CRPR) | 6-8 years
  Child social-relational risk factors, parent-report.
The Security Scale | 6-8 years
  To assess the child's perceptions of attachment security to their mother
Anthropometric Measures | 6-8 years
  weight, height, waist circumference, waist-to-hip ratio, waist-to-height ratio, head circumference and digit ratio (2D-4D).
Etch-a-Sketch Task | 6-8 years
  Parent-child interaction: video-recording of three joint parent-child activities (Etch-a-Sketch, block puzzles and a card game).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Dazzan, MD MSc PhD FRCPsych, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Study data will be analysed and results will be submitted for publication; participant identity will not be revealed. Study data will be retained and may be used in future studies, if this happens, further Research Ethics Committee approval will be sought.
  Authorised persons such as researchers, sponsors, regulatory authorities and Research and Development audit will have access to view identifiable data, for monitoring of the quality of the research.
  Study data will be retained for 20 years after completion of the study; and will be disposed of securely.